CLINICAL TRIAL: NCT02556515
Title: Total Joint Replacement or Interpositional Arthroplasty for the Treatment of Arthritis in the Carpometacarpal Joint of the Thumb
Brief Title: Joint Replacement or Interpositional Arthroplasty for CMC1 Arthritis, a Prospective Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Thorkildsen, Senior Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 276-08457c
Record Dates: First submitted 2014-02-17; First posted 2015-09-22 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthrosis of the Carpometacarpal Joint of the Thumb
Keywords: CMC1; arthritis; degenerative arthritis; thumb; interpositional arthroplasty; total joint replacement
MeSH Terms: conditions — Arthritis; Osteoarthritis | interventions — Arthroplasty, Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trapeziektomi and ligament interposition (Active Comparator): Interpositional arthroplasty Interpositional arthroplasty (Burton-Pellegrini procedure)
  Interventions: Procedure: Interpositional arthroplasty (Burton-Pellegrini procedure)
- Total joint replacement (Experimental): Elektra CMC1 uncemented prosthesis Elektra prosthesis
  Interventions: Procedure: Total joint replacement; Device: Elektra prosthesis

INTERVENTIONS:
Procedure: Interpositional arthroplasty (Burton-Pellegrini procedure) — Burton-Pellegrini procedure
  Arms: Trapeziektomi and ligament interposition
Procedure: Total joint replacement — Total joint replacement
  Other Names: Elektra prosthesis (Dijon, France)
  Arms: Total joint replacement
Device: Elektra prosthesis — Elektra prosthesis
  Arms: Total joint replacement

SUMMARY:
Interpositional arthroplasty is by many considered to be the current gold standard for the treatment of thumb carpometacarpal arthritis. The results are generally good, but the rehabilitation time can be long and failures are difficult to treat. Total joint replacements now exist with modern uncemented designs that can be an alternative treatment. Short term studies show that thumb function often is better and rehabilitation time shorter, however there is uncertainty with regards to the longevity of the implants. Currently no prospective randomized trials have compared these two treatment options. Our hypothesis is that the total joint replacement will give the same results or better when compared to the interpositional arthroplasty.

DETAILED DESCRIPTION:
Eligible: patients >18 years with pain and dysfunction from the first cmc joint. Clinical and radiological arthritis.

Exclusion: degenerative changes in the STT joint (all patients are assessed by CT), other injuries in the hand/thumb, pregnancy

Outcome measures: quick-Dash, Nelson hospital score, range of motion, grip strength

Complications are registered.

The patients are observed for two years and the investigators aim to include a total of 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* CMC 1 arthritis
* Pain and dysfunction
* Adult patients
* General good health

Exclusion Criteria:

* Pregnancy
* STT arthritis (CT scan preoperatively for all patients)
* Other injuries in thumb/hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11-24 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
quick-DASH | Baseline (preoperatively), and change from baseline postoperatively at 6 weeks, 3, 6, 12 and 24 months.
  two-page questionnaire with VAS-scale for pain and function.

SECONDARY OUTCOMES:
Nelson hospital score | Baseline (preoperatively) and change from base line postoperatively at 6 weeks, 3, 6, 12 and 24 months.
  one page thumb-specific questionnaire first published In Journal of Hand Surgery (Eur) 2007, 32E: 5: 524-528

OTHER OUTCOMES:
Grip strength | baseline (preoperatively) and change from base line postoperatively at 6 weeks, 3, 6, 12 and 24months
  Grip strength, key grip, tip-pinch measured by Jamar dynameter at each follow up
range of motion | baseline (preoperatively) and change from base line postoperatively at 6 weeks, 3, 6, 12 and 24 months
  Range of motion measured clinically (Kapandji opposition) and by x-ray (abduction, adduction, extension and flexion) at follow-up
complications | registered at 2 and 6 weeks. Thereafter at 3,6, 12 and 24 months.
  complications to either treatment form will be registered and published

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Thorkildsen, MBBS(Bsc), Principal Investigator — Hand- and microsurgical unit, Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No